CLINICAL TRIAL: NCT02676570
Title: Validation of Pathologic Diagnosis of Invasive Fungal Infection by Molecular Method - Retrospective Study Using Residual Storage Tissue Specimen
Brief Title: Validation of Pathologic Diagnosis of Invasive Fungal Infection by Molecular Method
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Dong-Gun Lee, Professor, Seoul St. Mary's Hospital
Other Study IDs: KC15SISI0338; IN-US-131-1971 (Other: Gilead ISR)
Record Dates: First submitted 2016-01-29; First posted 2016-02-08 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Mycoses
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Study specimen : Tissue Study content analysis: To determine fungal species and genetic mutations associated with drug resistance by extracting fungal DNA, but not patients' genetic information
Oversight: Data Monitoring Committee: No

SUMMARY:
1. Isolate fungal DNA(Deoxyribonucleic acid) from paraffin-fixed tissue specimens to distinguish and compare Aspergillus species to the existing optical pathological diagnosis.
2. PCR(polymerase chain reaction) validation.
3. Compare PCR results, microbial results and treatment results with the medical record.

DETAILED DESCRIPTION:
This study is a retrospective PCR(polymerase chain reaction) analysis of paraffin-fixed sample with a participants chart review. The PCR analysis will consist of two phases; a PCR test validation phase and an azole resistance test phase. The investigators will also perform a retrospective chart review to investigate the association of participants' fungal clinical outcomes and the presence of azole resistance.

I. PCR analysis

1. PCR test validation phase

   * Validating PCR assay by mock tissues and Invasive fungal infection proven tissues(microbiologically and pathologically proven cases).
   * The number of validation samples will be 1000 (200 samples * five target PCR).
   * For the enough validation of PCR results, inter-laboratory comparisons, especially with the core laboratory, are performed to verify the PCR results of the same test sample among laboratories and to standardize a certain protocol for the molecular identification of fungal infection from the clinical specimens.
   * Positive controls (human β-globin gene and mouse actin gene) and negative controls (non-infected samples) are used for validating of PCR assays. Precision of each PCR set is checked using the false discovery rate (FDR) which can be the acceptable level of false positives among a set of significant results. If FDR is >5%, it will be rejected.
   * The intra-assay repeatability will be evaluated on 10 replicates of one of the DNA subsamples analyzed in a single assay. The inter-assay reproducibility will be assess on the same DNA subsample five separate times while the inter-sample reproducibility will be determine on separate extractions of the four subsamples amplified a single time. Statistical analysis will be carry out using SAS software.
2. Azole resistance test phase

   * The investigator will perform a PCR assay using participants biopsied paraffin embedded tissues. Technical method of the PCR assay is attached separately.
   * Around a hundred biopsied samples under impression of fungal infection from June 1st, 2009 to June 31st, 2014 will be included for the PCR testing.

II. Retrospective chart review of all enrolled participants.

1. Data collection

   * All available participants' electronic medical record data will be reviewed for collecting demographic and clinical information.
2. Outcome measures

   * The investigators will evaluate Invasive fungal infecrion treatment results, survival rates, and prognosis according to the existence of azole resistance and antifungal treatment modalities including medications.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with invasive fungal disease based on the biopsy from June 2009 to May 2014

Exclusion Criteria:

* Patients who do not currently have residual paraffin-fixed specimens

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were diagnosed with invasive fungal disease based on the biopsy from June 2009 to May 2014
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Identify of fungal species by PCR method | two years
  Identify fungal DNA in Paraffine embedded tissue specimens. The outcome will be describe as success or fail

SECONDARY OUTCOMES:
Invasive fungal infection treatment success rate | two years
  Evaluate of Invasive fungal infection treatment success rate.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Gun Lee, M.D., Ph.D., Principal Investigator — Division of Infectious Diseases, Department of Internal Medicine, The Catholic Blood and Marrow Transplantation Center, Vaccine Bio Research Institute, College of Medicine, The Catholic University of Korea, Seoul, Korea

IPD SHARING:
Plan to Share IPD: No